CLINICAL TRIAL: NCT02249130
Title: Tipranavir (PNU-140690): A Fourteen Day Dose-response Study Using a Prototype Self-emulsifying Drug Delivery System (SEDDS) Formulation in Treatment-naive HIV-1 Infected Patients. Report on the Post-study Option, a 46-week Treatment Period of Triple Therapy With Delavirdine, ZDV and 3TC Without Tipranavir
Brief Title: Tipranavir Dose-response Study Using a Prototype Self-emulsifying Drug Delivery System (SEDDS) Formulation in Treatment-naive HIV-1 Infected Patients Report on the Post-study Option, a Treatment of Triple Therapy With Delavirdine, ZDV and 3TC Without Tipranavir
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1182.3
Record Dates: First submitted 2014-09-23; First posted 2014-09-25 (Estimated); Last update posted 2014-09-25 (Estimated); Status verified 2014-09

CONDITIONS: HIV Infections
MeSH Terms: conditions — HIV Infections | interventions — tipranavir; Ritonavir; Delavirdine; Zidovudine; Lamivudine; Stavudine

ARMS (1):
- Treatment of HIV- infected patients (Experimental): 14 days treatment with tipranavir, ritonavir, then 46 weeks of triple- treatment with delavirdine, zidovudine and lamivudine (stavudine for patients intolerant of zidovudine)
  Interventions: Drug: Tipranavir (TPV); Drug: Ritonavir (RTV); Drug: Delavirdine (DLV); Drug: Zidovudine (ZDV); Drug: Lamivudine (3TC); Drug: Stavudine (d4T)

INTERVENTIONS:
Drug: Tipranavir (TPV)
Drug: Ritonavir (RTV)
Drug: Delavirdine (DLV)
Drug: Zidovudine (ZDV)
Drug: Lamivudine (3TC)
Drug: Stavudine (d4T)

SUMMARY:
To investigate the safety of a standard triple therapy regimen of delavirdine (DLV), zidovudine (ZDV), and lamivudine (3TC) following 14 days of experimental treatment with regimens of tipranavir (TPV) with and without ritonavir (RTV)

ELIGIBILITY:
Inclusion Criteria:

* HIV-1 RNA ≥ 5,000 copies/mL by Roche Amplicor assay
* CD4 cell count ≥ 50 cells/mm3
* Karnofsky performance status ≥ 80
* Age ≥ 13 years
* Screening laboratory values indicative of adequate baseline organ function, Grade 0 or 1 for laboratory values based on the ACTG toxicity scale grade. Selected stable [2 months or longer] Grade 2 laboratory abnormalities were subject to sponsor's approval
* Acceptable medical history and physical examination
* Agreement to use a barrier contraceptive method for at least 1 month prior to the administration of the study medication, during the study, and for 30 days after the end of the study
* Signed informed consent
* To enter the post-study option, patients have to have completed the 14-day tipranavir phase of the trial

Exclusion Criteria:

* Previous treatment with any antiretroviral drugs for more than 2 weeks
* Clinically significant, active and/or acute (onset within the prior month) medical problems including opportunistic infections, such as active cryptococcosis, Pneumocystis carinii pneumonia (PCP), herpes zoster, histoplasmosis or cytomegalovirus (CMV) , or non-opportunistic diseases including, but not limited to, progressive multifocal leukoencephalopathy, lymphoma, or malignancy requiring systemic therapy
* History of clinically significant nervous system or muscle diseases, seizure disorder, or psychiatric disorder that might impair compliance with the study
* Receipt of any known enzyme-inducing drugs including rifabutin, rifampin, carbamazepine, dexamethasone, phenobarbital, phenytoin, sulfamidine, sulfinpyrazone, or troleandomycin within 30 days prior to participation in the study
* Receipt of any investigational medication within 30 days prior to participation in the study
* Receipt of oral contraceptives within 30 days prior to participation in the study
* Pregnancy or lactation (serum ß-human chorionic gonadotropin (ß-HCG) test negative at second screen visit of the tipranavir phase of trial)
* Evidence of active substance abuse that, in the investigator's opinion, could affect study adherence
* In the investigator's judgment, inability to comply with the protocol requirements for reasons other than those specified above

Min Age: 13 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 1999-03; Primary Completion 2000-04 (Actual)

PRIMARY OUTCOMES:
Number of patients with treatment-emergent adverse events | Up to 46 weeks
Number of patients with drug-related adverse events | Up to 46 weeks
Number of patients with AIDS clinical trials group (ACTG) grade 3 or 4 toxicity | Up to 46 weeks
Number of patients with a treatment toxicity leading to study discontinuation | Up to 46 weeks
Number of patients with serious treatment-emergent adverse events | Up to 46 weeks
Number of patients with changes in laboratory parameters | Up to 46 weeks
  Only lab values associated with metabolic disorders